CLINICAL TRIAL: NCT00525642
Title: A Chinese Multi-Center,Randomized Study of Combination or Sequential Use of Docetaxel,Anthracycline and Cyclophosphamide in Adjuvant Therapy for Node Positive Breast Cancer
Brief Title: Study of Suitable Schedule of Docetaxel,Anthracycline and Cyclophosphamide in Adjuvant Therapy of Beast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX-619
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2007-09-06 (Estimated); Status verified 2007-08

CONDITIONS: Breast Neoplasms; Adjuvant; Chemotherapy
Keywords: Breast-adjuvant; Breast-chemotherapy; Combination chemotherapy regimens
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): six cycles of adjuvant TAC
  Interventions: Drug: Docetaxel, Doxorubicin or Epirubicin, Cyclophosphamide
- B (Experimental): four cycles of T followed by 4 cycles of AC
  Interventions: Drug: Docetaxel, Doxorubicin or Epirubicin, Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel, Doxorubicin or Epirubicin, Cyclophosphamide — Docetaxel 75mg/m2, doxorubicin 50mg/m2 or epirubicin 60mg/m2, cyclophosphamide 500mg/m2 six cycles
  Other Names: Docetaxel=Taxotere®
  Arms: A
Drug: Docetaxel, Doxorubicin or Epirubicin, Cyclophosphamide — Docetaxel 100mg/m2 four cycles; Doxorubicin 60mg/m2 or epirubicin 75mg/m2 ,cyclophosphamide 600mg/m2) four cycles
  Other Names: Docetaxel= Taxotere®
  Arms: B

SUMMARY:
Anthracycline based regimens followed by a taxane (CALGB-9344 trial and NSABP-B28) or reversed (MD Anderson Adjuvant Trial) has already accepted as adjuvant therapy for node positive breast cancer. Also in this group of patients, data from BCIRG-001 trial had shown that six cycles of adjuvant TAC (docetaxel, doxorubicin and cyclophosphamide) is superior to standard FAC (5-FU, doxorubicin and cyclophosphamide ) combination in terms of both disease free and overall survival, while associated with a higher rate of febrile neutropenia. Then question arose whether it is better to use docetaxel and anthracycline in combination or sequence.

DETAILED DESCRIPTION:
In this national wide study, women with node positive operable breast cancer are eligible for inclusion.Patients were designed to randomize to six cycles of adjuvant TAC (Taxotere® 75mg/m2, doxorubicin 50mg/m2 or epirubicin 60mg/m2, cyclophosphamide 500mg/m2), and four cycles of T(100mg/m2), followed by 4 cycles of AC(doxorubicin 60mg/m2 or epirubicin 75mg/m2 ,cyclophosphamide 600mg/m2). Prophylaxis with G-CSF was allowed for two arms when febrile neutropenia occurred in the first cycle of the study treatment. The second endpoint of this study is disease free survival. The primary objective is to compare the disease free survival rate and safety profiles of the above mentioned two arms.

ELIGIBILITY:
Inclusion Criteria:

* pT1-3,pN1-3,M0, operable breast cancer
* Karnofsky >=80
* Pregnant test negative

Exclusion Criteria:

* Prior Chemotherapy with anthracyclines and / or Taxanes, except for Neoadjuvant therapy
* Prior breast radiation
* Bilateral breast cancer
* in-operable breast cancer
* Other health condition which may be contraindications for chemotherapy
* contraindications for Dexamethasone

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2003-06; Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years and 10 years
Grade III/IV Adverse Event,Severe Adverse Event | during chemotherapy and 30 days after treatment

SECONDARY OUTCOMES:
Overall Survival | 5 years and 10 years
Distant disease free Survival | 5 years and 10 years
Time to treatment failure | 5 years and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhou Shen, M.D., Study Chair — Cancer Hospital / Institute, Fudan University; Zhiming Shao, M.D., Study Director — Cancer Hospital / Institute, Fudan University
Locations (5):
- China (5):
  - Beijing 307 Hospital, Beijing, Beijing Municipality
  - No2 affiliated hospital of Sun Yat-sen medical Univesity, Guangzhou, Guangdong
  - Liaoning Province Cancer Hospital, Shenyang, Liaoning
  - Cancer Hospital / Institute, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai No.6 hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Yang L, Li LD, Chen YD, Parkin DM. [Time trends, estimates and projects for breast cancer incidence and mortality in China]. Zhonghua Zhong Liu Za Zhi. 2006 Jun;28(6):438-40. Chinese. PMID 17152490
- [Background] Martin M, Pienkowski T, Mackey J, Pawlicki M, Guastalla JP, Weaver C, Tomiak E, Al-Tweigeri T, Chap L, Juhos E, Guevin R, Howell A, Fornander T, Hainsworth J, Coleman R, Vinholes J, Modiano M, Pinter T, Tang SC, Colwell B, Prady C, Provencher L, Walde D, Rodriguez-Lescure A, Hugh J, Loret C, Rupin M, Blitz S, Jacobs P, Murawsky M, Riva A, Vogel C; Breast Cancer International Research Group 001 Investigators. Adjuvant docetaxel for node-positive breast cancer. N Engl J Med. 2005 Jun 2;352(22):2302-13. doi: 10.1056/NEJMoa043681. PMID 15930421
- [Background] Nabholtz JM, Falkson G, Campos D, et al. A phase III trial comparing doxorubicin (A) and docetaxel (T) (AT) to doxorubicin and cyclophosphamide (AC) as first line chemotherapy for MBC. Proc. Amer. Soc. Clin. Oncol. (1999) 18: 127a (Abstr 485).
- [Background] I.B.Ambulkaar, et al.Neoadjuvant sequential chemotherapy with docetaxel followed by epirubicin and cyclophosphamide in locally advanced breast cancer. Proc. Amer. Soc. Clin. Oncol. 2003 (Abstr 226)